CLINICAL TRIAL: NCT02891317
Title: Assessing Ocular Hemodynamic Response to Surgical Intervention in Glaucoma
Status: Terminated | Type: Observational
Why Stopped: Technical & Logistical issues
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Eye Institute (NEI) (NIH); American Glaucoma Society (Other)
Responsible Party: Sponsor
Other Study IDs: 14-3339; 1K23EY026098-01 (NIH)
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Primary Open Angle Glaucoma; Low Tension Glaucoma; Cataract; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma; Cataract; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cataract Surgery Only: Twenty-five participants with mild or moderate open angle glaucoma (OAG) controlled by medication with a visually significant cataract that meets clinical criteria for cataract surgery will be recruited from the glaucoma clinics at the UNC Kittner Eye Center. Patients who are consented for cataract surgery only (Group 1) will be recruited to this group. Each procedure will be completed in a standardized fashion with standardization of the post-operative medications. An effort will be made to gender and age match each surgical group as well as provide reasonable racial and ethnic diversity.
- Cataract Surgery with iStent: Twenty-five participants with mild or moderate open angle glaucoma (OAG) that meets clinical criteria for cataract surgery with implantation of an iStent trabecular micro-bypass shunt will be recruited from the glaucoma clinics at the UNC Kittner Eye Center. Patients who are consented for cataract surgery with iStent (Glaukos Corp., Laguna Hills, CA) implantation (Group 2) will be recruited to this group. Each procedure will be completed in a standardized fashion with standardization of the post-operative medications. An effort will be made to gender and age match each surgical group as well as provide reasonable racial and ethnic diversity.
- Glaucoma Drainage Device: Twenty-five participants with moderate or severe open angle glaucoma (OAG) that meets clinical criteria for implantation of a glaucoma drainage device (Group 3) will be recruited from the glaucoma clinics at the UNC Kittner Eye Center. Patients who are consented for implantation of a glaucoma drainage device (Group 3) will be recruited to this group. There will be 25 participants in each of the groups. Each procedure will be completed in a standardized fashion with standardization of the post-operative medications. An effort will be made to gender and age match each surgical group as well as provide reasonable racial and ethnic diversity.

SUMMARY:
The purpose of this study is to assess how surgical interventions in glaucoma affect 24-hour intraocular pressure, 24-hour ocular perfusion pressure, optic nerve blood flow, and retinal oxygen saturation.

DETAILED DESCRIPTION:
Purpose: Glaucoma is the leading cause of irreversible blindness worldwide and the third leading cause of vision loss in the United States. It is estimated that greater than 4.3 million Americans will have glaucoma in 2030. The treatment options are topical medications, laser surgery, and incisional surgery. The goal of therapy is to lower intraocular pressure (IOP). Despite adequate lowering of IOP, many patients continue to lose vision due to progressive glaucomatous optic atrophy. This is likely related to the poor understanding of glaucoma pathogenesis. There are two theories which explain the mechanism of primary open angle glaucoma (POAG). The mechanical theory posits that intraocular pressure (IOP) can produce optic nerve damage through biomechanical or structural factors. All current therapeutic interventions are aimed at this particular mechanism. The vascular theory suggests that compromise of the optic nerve microvasculature induces glaucomatous optic nerve damage. There is a significant body of literature supporting the role of ocular hemodynamic (OHD) changes in the development and progression of glaucoma. However, there have been limited investigations of the effect of surgical interventions on OHD. This is primarily due to a lack of non-invasive, cost-effective methods of assessing OHD factors. Today, the technology exists to assess these factors in such a manner. Thus, the purpose of this study is to assess the response of OHD factors to surgical intervention in glaucoma patients. Participants: Seventy-five participants with varying degrees of open angle glaucoma (OAG) that meet clinical criteria for cataract or glaucoma surgery will be recruited from the glaucoma clinics at the University of North Carolina (UNC) Kittner Eye Center. Once they have been determined to be eligible, they will be assigned to one of three groups based upon surgical indication. Group 1 is cataract surgery only. Group 2 is cataract surgery with iStent (Glaukos Corp., Laguna Hills, CA) implantation. Group 3 is implantation of a glaucoma drainage device. Each procedure will be completed in a standardized fashion with standardization of the post-operative medications. An effort will be made to gender and age match each surgical group as well as provide reasonable racial and ethnic diversity. Procedures (methods): Participants will undergo assessment of 24 hour IOP and ocular perfusion pressure (OPP), retinal oxygen saturation (RSO2), and optic nerve blood flow (ONBF), within 10 days of their assigned surgical procedure and again 6-8 weeks post-operatively. Ambulatory IOP and OPP: IOP will be measured using the Triggerfish® (Sensimed AG, Lausanne, Switzerland) contact lens sensor (CLS) every five minutes. Blood pressure (BP) will be measured with an ambulatory BP measure (ABPM) every 30 minutes during the day and every hour overnight. Participants will have the CLS and ABPM placed by study personnel, wear them for 24 hours assuming their typical daily activity and sleep regimen, then return to clinic the following day to have the devices removed. Optic Nerve Blood Flow and Retinal Oximetry: Prior to placement of the CLS and ABPM participants will undergo assessment of the ONBF using Doppler spectral domain optical coherence tomography (SD-OCT) and RSO2 using the Oxymap T1 (Oxymap, Reykjavik, Iceland) retinal oximeter.

ELIGIBILITY:
Inclusion Criteria:

* Participants meeting the following surgical indications for glaucoma:

  1. Open angle glaucoma with uncontrolled intraocular pressure on maximum tolerated medical therapy at risk of glaucomatous vision loss, documented visual field progression, severe visual field defects threatening or involving fixation with preserved visual acuity
  2. Phacomorphic angle closure with clinical symptoms and/or Visual Field/Optical Coherence Tomography defects
  3. Other appropriate indication
* Participants willing to complete the written informed consent
* Participants willing to complete a screening visit and subsequent study visits

Exclusion Criteria:

* Children and adolescents
* Patients with non-phacomorphic angle closure or secondary glaucoma diagnosis
* Prior retinal or glaucoma laser or incisional surgeries
* Non-glaucomatous optic neuropathy
* Any intraocular surgery within the preceding 90 days
* Active ocular infection or inflammation
* Ocular abnormalities that preclude the necessary study related measurements and assessments
* Pre-existing medical conditions that are associated with blood pressure (BP) instability
* Medications that confound BP assessment
* Symptomatic dry eye disease
* Allergy to silicone, adhesives, diagnostic and post-surgical topical ocular medications
* Skin irritation, eczema, or other indication against wearing patches
* Vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are clinically indicated and already scheduled to undergo one of the following surgical interventions: i) phacoemulsification with intraocular lens implantation, ii) phacoemulsification with intraocular lens and iStent implantation, and iii) glaucoma drainage device (GDD) implantation will be recruited from the glaucoma clinics of the University of North Carolina (UNC) Kittner Eye Center. Patients, 18 - 99, male and female, from every race and ethnicity will be recruited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Change in Intraocular Pressure | 7-10 days before surgery, 6-8 weeks post-operatively
  Trends in 24 hr IOP will be assessed using the Triggerfish contact lens system. Subjects will wear the lens on the surgical eye before and after surgery. Intraday and nocturnal trends will be analyzed. Additionally, ocular biometric measurements will be acquired and used in conjunction with the Triggerfish lens to develop a conversion factor for Triggerfish measurements (mV Eq) to intraocular pressure measurements (mmHg).

SECONDARY OUTCOMES:
Change in Optic Nerve Blood Flow | 7-10 days before surgery, 6-8 weeks post-operatively
  The trends of Doppler blood flow as measured with the Bioptigen Envisu C3500 will be assessed before and after surgery. Qualitative and quantitative analysis of flow velocities and capillary density will be completed.
Percent change in Retinal Oxygen Saturation | 7-10 days before surgery, 6-8 weeks post-operatively
  Retinal oxygen saturation will be assessed before and after surgery, glaucoma patients tend to have decreased oxygen utilization, thus higher venous O2 saturation. Data will be analyzed to determine whether tissue oxygen utilization improves with surgery.
Change in Ocular Perfusion Pressure | 7-10 days before surgery, 6-8 weeks post-operatively
  Ocular perfusion pressure (OPP) is the difference between the systemic blood pressure and the intraocular pressure. We will use measurements from an ambulatory blood pressure monitor and the Triggerfish lens to calculate OPP.

CONTACTS AND LOCATIONS:
Overall Officials: O'Rese J Knight, MD, Principal Investigator — Unverisity of North Carolina - Chapel Hill
Locations (1):
- UNC Kittner Eye Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No